CLINICAL TRIAL: NCT00533481
Title: Efficacy of MK0557 in Combination With Sibutramine or Orlistat (0557-015)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0557-015; 2007_615
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — spiro(cyclohexane-1,3'(1'H)-furo(3,4-C)pyridine)-4-carboxamide, N-(1-(2-fluorophenyl)-1h-pyrazol-3-yl)-1'-oxo-, trans-

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0557

SUMMARY:
Study medicine will be given alone, or in combination with either sibutramine or orlistat, to obese subjects to compare the effect on body weight over a six month period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-65 who are considered obese (have a body mass index between 30 and 43)

Exclusion Criteria:

* Subject has high blood pressure or is taking any high blood pressure medicine
* History of psychiatric disorder, stroke, or heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2004-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC